CLINICAL TRIAL: NCT05090527
Title: Penicillin Delabeling With Help of a Risk Stratification Tool, Advanced Provocation Tests in a Non Allergologic Unit
Brief Title: Penicillin Allergy Delabeling Project
Acronym: PenProv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Fonna (Other); Helse Forde (Other); Haraldsplass Deaconess Hospital (Other); Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 199210
Record Dates: First submitted 2021-08-09; First posted 2021-10-22 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-09

CONDITIONS: Penicillin Allergy
Keywords: penicillin allergy; clinical pathway; implementation; delabeling

STUDY DESIGN:
Intervention Model Description: Entry criteria: Penicillin allergy noted in patients journal or patient reported.
Masking Description: None, open provocation test with amoxicillin for eligible patients after risk stratification with a questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Directly delabeled trough risk stratification tool (Active Comparator): Patients who are stratified as " no penicillin allergy" undergo a one dose full dose provocation test with 500 mg amoxicillin.
  Interventions: Diagnostic Test: Risk stratification
- Low risk patients (Active Comparator): Patients stratified as low risk on penicillin provocation undergo a one dose full dose provocation test with 500mg amoxicillin
  Interventions: Diagnostic Test: Risk stratification
- High risk (Active Comparator): Patient stratified as high risk undergo a full allergologic work up, and only some of these will undergo a provocation test.
  Interventions: Diagnostic Test: Risk stratification

INTERVENTIONS:
Diagnostic Test: Risk stratification — advanced penicillin challenge after risk stratification

SUMMARY:
A investigational study to establish:

1. A validated cllinical pathway for delabeling declared Penicillin allergiy outside allergologic departments.
2. A survey to examine anesthesiologists attitudes and knowledge about penicillin delabeling.
3. A qualitative focus group study investigating barriers and facilitators in penicillin delabeling among hospital nurses and physichians.

2. Implement the pathway for delabeling declared penicillin allergy outside allergologic clinics across the Western Norway health region.

DETAILED DESCRIPTION:
Patients labeled penicillin allergic is a significant and growing public health problem. 10% of all patients report penicillin allergy. 9 out of 10 however tolerate penicillin on provocation, To be labeled as penicillin allergic has several well documented negative health outcomes for the individual, and on a public health scale.

One of the biggest obstacles in delabeling penicillin allergy is the lack of validated tools i Norwegian, the lack of in vitro tests for severe late /T cell mediated reactions and the accessibility of the gold standard procedure, drug provocation test.

In this study patients having a penicillin allergy label will after giving their written concent be screened used a risk stratification tool. The low risk patient will then directly undergo a single full dose amoxicillin challenge. High risk patients are refered to a allergologic clinic and undergoes full allergologic examination. The investigators seek to document that in low risk patients is a single dose Amoxicillin challenge safe and beneficial outside an allergologic clinic, and to validate the risk stratification tool in Norwegian.

To implement such pathways i qualitative data is needed to facilitate the right efforts and translate the method into every day clinical practice in a sustainable way. Here a anesthesiologist survey and focus group interviews with hospital nurses and physichians is planned.

Finally we will implement the method in an implementation study across the Western Norway Health region

ELIGIBILITY:
Inclusion Criteria:

* Penicillin allergy in the patient journal oder patient reported

Exclusion Criteria:

* Not able to give concent. Under 16 years of age.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Validating of a risk stratification tool ( in Norwegian) and advanced drug provocation challenge | 24 months
  Negative predictive value of the risk stratification tool

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events on oral provocation testing. | 24 months
  number of patients with treatment related adverse event on oral provocation testing.
Number of patients correctly delabeled | 24 months
  Og the patientents included in the implementation in clinical practice, how many had a correct procedure and result.

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir Storaas, phd, Study Chair — RAAO vest
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Helse Førde, Førde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alnaes MB, Oppegaard O, Kittang BR, Lygre SHL, Langeland AB, Skodvin B, Bjanes T, Storaas T. A new pathway for penicillin delabeling in Norway. World Allergy Organ J. 2023 Oct 16;16(11):100829. doi: 10.1016/j.waojou.2023.100829. eCollection 2023 Nov. PMID 37868111